CLINICAL TRIAL: NCT01230164
Title: Comparison of Four Different Aberrometers for Evaluation of Higher Order Visual Aberrations
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Other Study IDs: 09-03-016
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Normal Individuals With Visual Aberrations

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An aberrometer measures visual aberrations by mapping how light rays travel through the eye and by providing maps using colored gradients to represent the magnitude of refractive errors of the eye.

The purpose of this study is to compare 4 different aberrometers -Wavescan (Visx Technology), Zywave (Bausch & Lomb), Ladarwave aberrometer (Alcon Inc.) and Allegro Analyzer (Alcon Inc). In particular, the investigators propose to focus on the ability of these devices to display the higher order visual aberrations and to compare the quality of outputs from these 4 devices in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* male or female, at least 18 years of age
* no ocular abnormality other than refractive error
* patient in generally good & stable overall health
* has not worn contact lenses (hard or gas permeable lenses for at least 3 weeks and soft lenses for at least 3 days) prior to the study exam
* corneal topography must be normal, as judged by the investigator
* topical anesthesia and mydriatics must be tolerated
* patient must be able to fixate steadily
* ability to understand and provide informed consent to participate in this study

Exclusion Criteria:

* history of ocular surgery
* history of ocular trauma, infection, disease, or abnormality other than refractive error
* myopia or hyperopia > 7.0 D, astigmatism >3.0 D
* uncorrectable visual acuity below 20/20
* abnormal corneal topography pattern including, but not limited to keratoconus, forme fruste keratoconus, or corneal warpage
* pupil sizes below 6.0 mm under mydriasis
* iris problems including, but not limited to, coloboma and previous iris surgery
* ocular media problems, corneal, lens and/or vitreous opacities including, but not limited to cataract
* ocular movement abnormalities including, but not limited to, strabismus or nystagmus
* phenol red thread test (Zone Quick-Menicon Ltd) less than 9 mm/15 seconds
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects over the age of 18 with visual abberations.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pineda, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States